CLINICAL TRIAL: NCT05386563
Title: The Effect of Transcutaneous Auricular Vagal Nerve Stimulation (taVNS) on Pupillary Response and Perceptual Learning
Brief Title: taVNS on Pupillary Response and Perceptual Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 22-00516
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pupillary Response

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcutaneous Auricular Vagal Nerve Stimulation (taVNS) (Experimental)
  Interventions: Procedure: Transcutaneous Auricular Vagal Nerve Stimulation (taVNS)
- Sham (Sham Comparator)
  Interventions: Procedure: Sham Stimulation
- No Intervention (Control) (No Intervention)

INTERVENTIONS:
Procedure: Transcutaneous Auricular Vagal Nerve Stimulation (taVNS) — taVNS will be delivered by Digitimer DS7 Constant Current Stimulator (an FDA cleared medical device intended for human nerve and muscle stimulation).
  Stimulation is delivered via sticky pad electrodes all placed on the left side of the body (cymba concha, earlobe, and ulnar side of the wrist). Stimulation is delivered by a 3000ms pulse train (100us pulse width and 25Hz stimulation frequency). The current applied will be between 0.01uA to 9uA. The intervention will be delivered over the course of four sessions approximately one week apart.
  Arms: Transcutaneous Auricular Vagal Nerve Stimulation (taVNS)
Procedure: Sham Stimulation — Sham stimulation will be delivered by Digitimer DS7 Constant Current Stimulator (an FDA cleared medical device intended for human nerve and muscle stimulation).
  Stimulation is delivered via sticky pad electrodes all placed on the left side of the body (either earlobe or forearm).
  Arms: Sham

SUMMARY:
This study has two parts. The study team will evaluate transcutaneous auricular vagal nerve stimulation (taVNS) and two sham settings during a passive task while measuring pupillary response. Second, the study team will assign either taVNS, sham, or no intervention during a go/no-go task and evaluate perceptual learning over three sessions which will also include measuring the pupillary response and electroencephalogram (EEG).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals 18 to 65
* Normal audiometric testing

Exclusion Criteria:

* Co-morbidities including cardiomyopathies, arrhythmias
* Implantable devices including vagal stimulators, pacemakers
* Presence of metallic implants
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Change in Time It Takes to Reach 90% of Asymptotic Level Performance | Baseline, Month 3
  Will be measured during performance on a go/no-go task.
Change in Overall Mean Peak (Pupillary Response) | Baseline, Month 3
  Pupillary responses will be measured noninvasively using a video camera during a go/no-go task.
Change in Speed of Learning to Perform a Behavioral Task | Baseline, Month 3
  Will be measured during performance on a go/no-go task.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Svirsky, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health - Bellevue Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Researchers who provide a methodologically sound proposal will have access to the data upon reasonable request. Requests should be directed to mario.svirsky@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.